CLINICAL TRIAL: NCT01820182
Title: Prospective Comparison of the Diagnostic Yield of Small Bowel Pillcam SB2 and Capsocam Capsule in Patients With Obscure Digestive Bleedings
Brief Title: Prospective Comparison of the Diagnostic Yield of Small Bowel Pillcam SB2 and Capsocam Capsule
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Edouard Herriot (Other)
Collaborators: Capso Vision, Inc. (Industry)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Proffessor, Hôpital Edouard Herriot
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010-023341-29
Record Dates: First submitted 2013-03-21; First posted 2013-03-28 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Anemia; Gastrointestinal Bleedings; Méléna; Angiodysplasia; Polyps
MeSH Terms: conditions — Anemia; Angiodysplasia; Polyps | interventions — Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- capsocam capsula (Experimental): capsocam capsula readings
  Interventions: Device: capsule endoscopies

INTERVENTIONS:
Device: capsule endoscopies — Patients inclusion following inclusion criterias Randomization of capsule ingestion order Videocapsule recording by the two capsules Reading of the two capsules films in randomized order by two different readers in each center Reviewing of discordant capsule films by an expert panel
  Other Names: Pillcam SB2; Capsocam

SUMMARY:
Comparative, randomized study patients are scheduled to have two capsule endoscopies within 2 to 14 days from each other using two different endoscopies the Pillcam SB2 (Given Imaging, Israel) and the Capsocam (Capso Vision Saratoga United States) The order in which the devices are administered is randomly allocated.

DETAILED DESCRIPTION:
Objectives

Main objective

To compare the diagnostic yield of both capsules in the same patients with a satisfying concordance coefficient k>0,6

Secondary objectives

To compare the sensitivity and specificity of both capsule readings To copmpare the sensitivity and specificity for specific lesions classified in terms of relevance P0 P1 P2 To check the tecnical fiability (incidence of technical issues To check the feasibility To evaluate the rate of complete small bowel examination, the small bowel transit time the capsule reading time

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* obscure digestive bleeding justifying capsule endoscopy
* complete endoscopic work up including colonoscopy with ileoscopy and gastroscopy with aneathesia or sedation
* absence of concomittent ongoing study
* absence of occlusive symptoms of suspected Crohn's disease nor of previous small bowel radiotherapy
* filled inform consent
* no implanted pace maker
* patient being affiliated to the CPAM

Exclusion Criteria:

* under 18 years old
* oral iron within 8 days before capsule endoscopy
* gastroparesis
* pacemaker
* swallowing troubles
* presence of oclusive symptoms suspected Crohn's disease nor of previous small bowel radiotherapy
* pregnancy or risk of pregnancy without efficient oral contraception
* absence of written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
number of discordant films between the two capsules with two different readers | 14 days
  Reading of the two capsules film is randomized order by two different readers in each center

CONTACTS AND LOCATIONS:
Overall Officials: Saurin JS Jean Christophe, Msd, Principal Investigator

IPD SHARING:
Plan to Share IPD: No